CLINICAL TRIAL: NCT00369616
Title: Evaluation of Efficacy and Safety of Nicotine-Qbeta (NicQb) Vaccine Versus Placebo in Healthy Smokers
Brief Title: Efficacy and Safety of Nicotine-Qbeta Vaccine in Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT002-NicQb 02
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2008-03

CONDITIONS: Smokers
MeSH Terms: interventions — nicotine Qbeta vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- NicQb vaccine (Experimental)
  Interventions: Biological: CYT002-NicQb
- Placebo vaccine (Placebo Comparator)
  Interventions: Biological: CYT002-NicQb

INTERVENTIONS:
Biological: CYT002-NicQb

SUMMARY:
The purpose of this study is to help smokers quitting by vaccinating them with CYT002-NicQb. Upon vaccination, the smoker will generate antibodies directed against free nicotine. The antibodies will bind nicotine and prevent its passage into the brain. The successfully vaccinated smoker will have no reward effect after smoking, thus braking the vicious circle of nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 to 70 years
* Smokers: > 10 and ≤ 40 cigarettes per day and smoking history of more than 3 years
* Fageström Test for Nicotine Dependence (FTND) score ≥ 5
* Female participant must meet one of the following criteria: a) no reproductive potential due to menopause, hysterectomy, bilateral oophorectomy, or tubal ligation; b) agrees to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 12 additional months after the last immunization

Exclusion Criteria:

* Pregnant or nursing
* History of severe allergy or immunological disorders
* Blood donation within previous 30 days
* Surgery within previous 30 days
* Use of investigational drugs within previous 60 days
* Significant cardiovascular disease:

  * angina pectoris
  * congestive heart failure
  * clinically significant murmurs
  * previous angioplasty or coronary artery bypass surgery
* Active infectious disease:

  * WBC > 12 000 cells/µL
  * Seropositivity for Hepatitis B and C
  * History of risk behavior to acquire HIV
* Significant hepatic disease
* Significant renal disease
* Significant hematological disorder
* Significant pulmonary disease
* History of malignancy
* Autoimmune disease
* Organic neurological disorder or significant psychiatric disorder
* Use of psychoactive drug within one month before enrolment
* Abuse of drugs or alcohol
* Subjects using any concomitant medications due to chronic illness which bears a high risk of fluctuation in disease activity or exacerbations during a 12-months period such as coronary heart disease, asthma, severe COPD, chronic rheumatoid disease, diabetes, etc. should be excluded.
* Obesity: BMI > 35 kg/m2
* Use of concomitant nicotine replacement treatment (NRT) at screening or visit 1
* Any planned surgical intervention during the study period

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Abstinence from smoking defined as self-reported abstinence and confirmed by measurement of carbon monoxide in exhaled air less than 10ppm | Monthly up to month 6, and during follow-up at months 9 and 12
Immunogenicity of the vaccine, by measuring specific anti-nicotine IgG antibodies by ELISA | Baseline, monthly up to month 6, and months 9 and 12
Safety and tolerability by recording adverse events, injection site examinations, vital signs, standard clinical laboratory (serum chemistry, hematology) | Baseline, and at various times up to month 12

SECONDARY OUTCOMES:
Craving and withdrawal symptoms by Questionnaire on Smoking Urges and Wisconsin Withdrawal Scale | Baseline, monthly up to month 6

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Cornuz, Prof., Study Chair — Department of Medicine; University Hospital Lausanne, Switzeland; Thomas Cerny, Prof., Principal Investigator — Department of Medicine, Kantonsspital St. Gallen, Switzerland; Felix Jungi, MD, Principal Investigator — Department of Medicine, Kantonsspital St. Gallen, Switzerland; Karl Klingler, MD, Principal Investigator — Lung Center Hirslanden, Zuerich, Switzerland
Locations (3):
- Switzerland (3):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Lausanne (CHUV), Lausanne, Canton of Vaud
  - Lungenzentrum Hirslandenklinik Zuerich, Zurich, Canton of Zurich

REFERENCES:
- [Derived] Cornuz J, Zwahlen S, Jungi WF, Osterwalder J, Klingler K, van Melle G, Bangala Y, Guessous I, Muller P, Willers J, Maurer P, Bachmann MF, Cerny T. A vaccine against nicotine for smoking cessation: a randomized controlled trial. PLoS One. 2008 Jun 25;3(6):e2547. doi: 10.1371/journal.pone.0002547. PMID 18575629